CLINICAL TRIAL: NCT06028581
Title: The Effect of Breastfeeding Support System in Newborns on Developmental Findings and Discharge Time
Brief Title: The Effect of Breastfeeding Support System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Fatma GUL CAN, Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: AICU-GULCAN002
Record Dates: First submitted 2023-07-24; First posted 2023-09-08 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Breastfeeding support system will be applied to newborn babies in addition to breast milk.
  Interventions: Other: breastfeeding support system
- Control Group (No Intervention): Newborn babies will receive breast milk.

INTERVENTIONS:
Other: breastfeeding support system — Using the breastfeeding support system
  Arms: Experimental Group

SUMMARY:
It is aimed to determine the effect of breastfeeding support system applied in newborns on developmental findings and discharge time.The research was planned as an experimental study with experimental and control groups. The population of the study consisted of babies who received care and treatment in Iğdır State Hospital Neonatal Intensive Care Clinic between February and June 2023. The sample of the study was calculated using the G*Power computer program. In the calculation made, it was found that a total of 70 children, 35 of each for the control and experimental groups, should be included. In this study, the experimental group consisted of 36 children and the control group consisted of 35 children. Children selected by simple random sampling method were divided into groups by randomization and which group would be the experimental group and which group would be the control group were determined by randomization. Masking was done during data collection and data analysis. The data is in the analysis stage.

DETAILED DESCRIPTION:
Breast milk is a natural food with high bioavailability, easy to digest, which reduces the morbidity and mortality of the newborn, contains all the fluid, energy and nutrients necessary for physical, spiritual and mental development.Breastfeeding has a biological and emotional impact on mother and baby, has many immunological, psychological, social and economic benefits for both mother and baby, and is the best method for maternal health and healthy growth and development of infants.The bond between mother and baby after birth In the sensitive period in which successful breastfeeding will be established by establishing a new hospital, some babies need to be hospitalized in the neonatal intensive care unit (NICU) for various reasons. During hospitalization, mothers cannot be with their babies during all feedings and often have to empty their breasts with a pump. The pump does not have the same physiological effect as breastfeeding on the milk injection response.

Due to some problems arising from the breast or the baby, the baby may have problems in grasping and holding the breast. In such cases, a breastfeeding support system can be used.

The breastfeeding support system is based on the logic of stimulating the formation of prolactin by the baby's sucking of the milk, assuming that it comes from the breast, with the help of a plastic tube (usually a nasogastric tube) that is fixed to the breast on one end and the other end inside the bottle/container containing breast milk or formula.With this method, it is aimed to increase milk production and restart breastfeeding through active sucking of the newborn and stimulation of the breasts.

ELIGIBILITY:
1. Inclusion Criteria: Before age of 28 days
2. Exclusion Criteria: After age of 29 days

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
LATCH Breastfeeding Diagnostic Measurement Tool | After each breastfeeding an average of 4 days
  LATCH Breastfeeding Diagnostic Measurement The tool was developed by Jensen and Wallace in 1993 in Oregon. LATCH is a diagnostic tool created by analogy with the APGAR scoring system in terms of scoring method. Each item is evaluated between 0-2 points. The lowest 0 points and the highest 10 points are obtained from the scale. The Cronbach alpha coefficient of the LATCH Breastfeeding Diagnostic Measurement Tool was reported as 0.94 by Demirhan, 0.96 by Koyun, and 0.95 by Yenal and Okumuş.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma GUL CAN, PhD, Principal Investigator — Agri Ibrahim Cecen University; Eda GÜLBETEKİN, PhD, Principal Investigator — Igdir University; Selahattin KARAGÖZ KARAGÖZ, PhD, Principal Investigator — Iğdır State Hospital
Locations (1):
- Agri Ibrahim Cecen University, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No